CLINICAL TRIAL: NCT02448043
Title: Cutaneous Prostaglandin Application: Nail Growth, Nail Brittleness, and Eye Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, David Palmer, Assistant Professor of Clinical Ophthalmology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00200526
Record Dates: First submitted 2015-05-04; First posted 2015-05-19 (Estimated); Results first posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-11

CONDITIONS: Nail Growth Cessation; Intraocular Pressure
Keywords: brittleness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Right Hand Bimatoprost 0.01% drops, Left Hand Placebo (Other): * Bimatoprost 0.01% drops placed on the proximal nail folds of the right hand digits two times per day for 30 days.
  * Saline solution drops placed on the proximal nail folds of the left hand digits two times per day for 30 days.
  Interventions: Drug: Bimatoprost 0.01%; Other: Placebo: saline
- Left Hand Bimatoprost 0.01% drops, Right Hand Placebo (Other): * Bimatoprost 0.01% drops placed on the proximal nail folds of the left hand digits two times per day for 30 days.
  * Saline solution drops placed on the proximal nail folds of the right hand digits two times per day for 30 days.
  Interventions: Drug: Bimatoprost 0.01%; Other: Placebo: saline

INTERVENTIONS:
Drug: Bimatoprost 0.01% — Bimatoprost drops added to the proximal nail folds of the randomized study hand digits two times per day for 30 days
  Other Names: Lumigan 0.01%
Other: Placebo: saline — Placebo drops added to the proximal nail folds of the hand digits opposite the study hand two times per day for 30 days

SUMMARY:
Topical prostaglandin agents are used to help reduce eye pressure in glaucoma patients. Bimatoprost (Lumigan 0.01%) is such an agent (Allergan, Inc.). Several of our patients on bimatoprost and an observational study of patients on bimatoprost in another center reported that fingernails grew longer and became less brittle using the topical eye drops to the eyes. The purpose of the double-blinded study is to determine whether the application of the eye drops directly to the proximal nail fold of one hand using the opposite hand as a control will result in longer nails, less brittle nails, and reduced eye pressures should any of the medication be absorbed into the systemic circulation.

DETAILED DESCRIPTION:
In addition to our observations with topical bimatoprost on fingernail growth, Wand and colleagues applied bimatoprost to the base of the fingernails demonstrating a 16.9% increase in fingernail growth from baseline, and a 10.4% increase from baseline on untreated nail beds. Other than these two reports, there are no studies addressing this topic to our knowledge based on a Medline search for off-label use of this drug. Other relevant studies have addressed increased hair and eyelash growth with the prostaglandin agents. Researching the biochemistry of the relationship of prostaglandins to hair and nail growth, the final common pathway appears to be with protein kinase C and the production of tropocollagens. The dermatology literature has demonstrated that both hair and nail keratocytes reside in the nail bed suggesting that increased collagen production may enhance the growth of both the nail bed and nail plate, possibly reducing nail brittleness.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Normotensive or glaucoma suspects on no ocular medications
* No manicure within 2 weeks of the study.

Exclusion Criteria:

* Individuals on topical or systemic essential fatty acids (EFA's) in hand lotions, creams, ointments, or medication, or on biotin.
* Digits with signs of nail injury, deformity, or infection.
* Nail biters, nail polishers, artificial nail wear or gels, and nail and trimming and filing until the study endpoint.
* Women of childbearing age who are pregnant or who are trying to become pregnant.
* Individuals with allergies or sensitivity to prostaglandin agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-06-04 (Actual); Primary Completion 2016-05-06 (Actual); Study Completion 2016-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Palmer, MD, Principal Investigator — Northwestern University
Locations (1):
- David J. Palmer, MD, Glenview, Illinois, United States

REFERENCES:
- [Background] Weston BC. Migraine headache associated with latanoprost. Arch Ophthalmol. 2001 Feb;119(2):300-1. No abstract available. PMID 11176999
- [Background] Ziboh VA, Miller CC. Essential fatty acids and polyunsaturated fatty acids: significance in cutaneous biology. Annu Rev Nutr. 1990;10:433-50. doi: 10.1146/annurev.nu.10.070190.002245. No abstract available. PMID 2200473
- [Result] Khouri AS, Fechtner RD, Zimmerman, TJ. Latanoprost: A New Approach to the Treatment of Glaucoma. Today's Therapeutic Trends 14: 225-240, 1997
- [Result] Woodward DF, Krauss AH, Chen J, Lai RK, Spada CS, Burk RM, Andrews SW, Shi L, Liang Y, Kedzie KM, Chen R, Gil DW, Kharlamb A, Archeampong A, Ling J, Madhu C, Ni J, Rix P, Usansky J, Usansky H, Weber A, Welty D, Yang W, Tang-Liu DD, Garst ME, Brar B, Wheeler LA, Kaplan LJ. The pharmacology of bimatoprost (Lumigan). Surv Ophthalmol. 2001 May;45 Suppl 4:S337-45. doi: 10.1016/s0039-6257(01)00224-7. PMID 11434936
- [Result] Bean GW, Camras CB. Commercially available prostaglandin analogs for the reduction of intraocular pressure: similarities and differences. Surv Ophthalmol. 2008 Nov;53 Suppl1:S69-84. doi: 10.1016/j.survophthal.2008.08.012. PMID 19038626
- [Result] Sjoquist B. Human pharmacokinetic studies summary. Pharmacia and Upjohn Company Technical Report 9500155. March 25, 1995.
- [Result] Tan J, Berke S. Latanoprost-induced prostaglandin-associated periorbitopathy. Optom Vis Sci. 2013 Sep;90(9):e245-7; discussion 1029. doi: 10.1097/OPX.0b013e31829d8dd7. PMID 23912967
- [Result] Wand M, Shields BM. Cystoid macular edema in the era of ocular hypotensive lipids. Am J Ophthalmol. 2002 Mar;133(3):393-7. doi: 10.1016/s0002-9394(01)01412-x. PMID 11915838
- [Result] Cohen JL. Enhancing the growth of natural eyelashes: the mechanism of bimatoprost-induced eyelash growth. Dermatol Surg. 2010 Sep;36(9):1361-71. doi: 10.1111/j.1524-4725.2010.01522.x. PMID 20384750
- [Result] Johnstone MA. Hypertrichosis and increased pigmentation of eyelashes and adjacent hair in the region of the ipsilateral eyelids of patients treated with unilateral topical latanoprost. Am J Ophthalmol. 1997 Oct;124(4):544-7. doi: 10.1016/s0002-9394(14)70870-0. PMID 9323945
- [Result] Wand M. New side effect of Prostaglandins. Agsocietynet@aaoforums.aao.org. Jan 2015.
- [Result] Seed Oils and Essential Fatty Acids. Retrieved 5/21/12 http://www.naturopathica.com/system/user_files/attachments/7/original/Naturopathica_Seed_Oils.pdf
- [Result] Janis J (ed). Nail bed injuries. Essential of Plastic Surgery: A UT Southwestern Medical Center Handbook. St Louis, MO: Quality Medical Publishing, Inc: 560-567, 2007.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited voluntarily from private office practices (DP and AS), and a university-based practice (AT).
Period: Overall Study
Arm/Group | Right Hand Bimatoprost 0.01% Drops, Left Hand Placebo | Left Hand Bimatoprost 0.01% Drops, Right Hand Placebo
Started | 23 | 22
Completed | 20 | 18
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Protocol Violation | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Right Hand Bimatoprost 0.01% Drops, Left Hand Placebo | Left Hand Bimatoprost 0.01% Drops, Right Hand Placebo | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] — Range from 24-88 years of age Population: Number analyzed for each row differs from the Overall analyzed number because the 'All Participants', 'Male', and 'Female' rows identify different populations
  Years
    All participants | 60.30 (9.27) | 63.33 (15.26) | 61.61 (12.27)
    Male: number analyzed (Participants) | 2 | 1 | 3
    Male | 67 (7.07) | 88 (0) | 74 (13.11)
    Female: number analyzed (Participants) | 18 | 17 | 35
    Female | 59.28 (9.19) | 61.88 (14.39) | 60.5 (11.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 15 | 17 | 32
  Hispanic | 1 | 0 | 1
  Asian | 2 | 1 | 3
  Black | 2 | 0 | 2
Nail Length of Hands [Mean (Standard Deviation); unit: mm] | 12.5 (1.32) | 12.21 (1.74) | 12.39 (1.51)
Nail Length of Digits [Mean (Standard Deviation); unit: mm] — Population: In the "Left Hand Bimatoprost, Right Hand Placebo" group, 1 subject is missing a forefinger
  mm
    Thumb | 14.50 (1.68) | 13.85 (2.10) | 14.18 (0.30)
    Forefinger: number analyzed (Participants) | 20 | 17 | 37
    Forefinger | 12.26 (1.64) | 12.28 (1.94) | 12.27 (0.21)
    Middle Finger | 12.81 (1.70) | 12.52 (2.08) | 12.67 (0.27)
    Ring Finger | 12.50 (1.60) | 12.21 (2.04) | 12.35 (0.31)
    Pinky Finger | 10.42 (1.43) | 10.26 (1.66) | 10.34 (0.16)
Intraocular Pressure [Mean (Standard Deviation); unit: mm Hg] — Population: No baseline IOP data on 13 subjects
  mm Hg
    Both eyes: number analyzed (Participants) | 13 | 12 | 25
    Both eyes | 16.23 (3.85) | 13.67 (2.91) | 15 (3.64)
    Right eye: number analyzed (Participants) | 13 | 12 | 25
    Right eye | 16.00 (2.89) | 13.83 (3.24) | 14.96 (3.19)
    Left eye: number analyzed (Participants) | 13 | 12 | 25
    Left eye | 16.46 (4.74) | 13.5 (2.68) | 15.04 (4.10)
Nail Brittleness [Mean (Standard Deviation); unit: Score on a scale] — Scale Title: Nail Brittleness (1-4)
  Subjective assessment by subjects on scale of 1 (no brittleness) to 4 (maximum brittleness). Population: No or incomplete data 2 participants
  Score on a scale
    number analyzed (Participants) | 18 | 18 | 36
    (all) | 2.61 (0.98) | 2.42 (1.06) | 2.51 (1.01)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Nail Length of Hands
Description: Measured by digital calipers (Ironton 6 in. Stainless Steel Digital Fractional Caliper, Northern Tool and Equipment, Burnsville, MN, USA)
Time Frame: Baseline, 30 days
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Hands
Groups:
- Bimatoprost 0.01% Drops: Bimatoprost 0.01%: Bimatoprost drops added to the proximal nail folds of the randomized study hand digits two times per day for 30 days
- Placebo: Saline solution drops placed on the proximal nail folds of the hand digits opposite from the study hand two times per day for 30 days.
Arm/Group | Bimatoprost 0.01% Drops | Placebo
Number analyzed (Participants) | 38 | 38
Number analyzed (Hands) | 38 | 38
mm
  Total Nail Growth (power = 1.0) | 13.49 (1.14) | 15.10 (1.29)
  Individual Nail Growth | 1.34 (0.33) | 1.51 (0.48)
Statistical Analysis 1: Comparison: Bimatoprost 0.01% Drops vs Placebo; Test type: Superiority; p = 0.532, t-test, 2 sided — Threshold is p<0.05

2. Primary Outcome: Change From Baseline in Nail Length of Digits
Description: as for outcome 1
Time Frame: Baseline, 30 Days
Population: Excluding the negative growth nails and chipped nails combined; one subject is missing a forefinger
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Digits
Arm/Group | Bimatoprost 0.01% Drops | Placebo
Number analyzed (Participants) | 38 | 38
Number analyzed (Digits) | 189 | 190
mm
  Thumb: number analyzed (Digits) | 38 | 38
  Thumb | 1.58 (1.70) | 1.48 (1.82)
  Forefinger: number analyzed (Digits) | 37 | 38
  Forefinger | 1.26 (1.38) | 1.02 (2.76)
  Middle Finger: number analyzed (Digits) | 38 | 38
  Middle Finger | 0.90 (1.76) | 1.40 (1.50)
  Ring Finger: number analyzed (Digits) | 38 | 38
  Ring Finger | 1.33 (1.27) | 1.76 (1.77)
  Pinky Finger: number analyzed (Digits) | 38 | 38
  Pinky Finger | 1.63 (1.55) | 1.62 (1.65)
Statistical Analysis 1: Comparison: Bimatoprost 0.01% Drops vs Placebo; Test type: Superiority; p = 0.523, t-test, 2 sided — Threshold is p<0.05

3. Primary Outcome: Intraocular Pressure at 30 Days of Treatment
Description: IOP using a Goldmann applanation tonometer (GAT) between 7:30 AM and 10:00 AM
Time Frame: Between 7:30 AM and 10:00 AM at 30 days post treatment
Population: No IOP data on 13 subjects Missing final IOP data on 1 subject
  Arms are not grouped as 'Bimatoprost 0.01%' and 'Placebo' because this is a split-person study, so every participant received both the treatment and the placebo. Since this outcome is measuring eye pressure, there is no way to distinguish which group/arm is influencing eye pressure.
Measure: Mean (Standard Deviation); unit: mm Hg
Units Other Than Participants: Eyes
Arm/Group | Right Hand Bimatoprost 0.01% Drops, Left Hand Placebo | Left Hand Bimatoprost 0.01% Drops, Right Hand Placebo
Number analyzed (Participants) | 13 | 11
Number analyzed (Eyes) | 26 | 22
mm Hg
  Both eyes | 16.42 (3.24) | 13.91 (1.80)
  Right eye: number analyzed (Eyes) | 13 | 11
  Right eye | 16.38 (3.73) | 14.0 (2.10)
  Left eye: number analyzed (Eyes) | 13 | 11
  Left eye | 16.46 (2.82) | 13.82 (1.54)
Statistical Analysis 1: Comparison: Right Hand Bimatoprost 0.01% Drops, Left Hand Placebo vs Left Hand Bimatoprost 0.01% Drops, Right Hand Placebo; Comparing baseline values of both arms to completion values of both arms; Test type: Superiority; p = 0.912, t-test, 2 sided — Threshold is p<0.05

4. Primary Outcome: Nail Brittleness at 30 Days of Treatment
Description: Scale Title: Nail Brittleness (1-4)
  Subjective assessment by subjects on scale of 1 (no brittleness) to 4 (maximum brittleness).
Time Frame: Baseline, 30 days
Population: No or incomplete data on seven subjects
  Subjects were asked to assess nail brittleness of both hands and rank them together - i.e. the value each subject gave for nail brittleness was the combination of the placebo hand and the treatment hand. Nail brittleness values were not distinguished between the placebo hands and the treatment hands.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Right Hand Bimatoprost 0.01% Drops, Left Hand Placebo | Left Hand Bimatoprost 0.01% Drops, Right Hand Placebo
Number analyzed (Participants) | 16 | 15
Score on a scale | 2.25 (0.93) | 2.43 (1.10)
Statistical Analysis 1: Comparison: Right Hand Bimatoprost 0.01% Drops, Left Hand Placebo vs Left Hand Bimatoprost 0.01% Drops, Right Hand Placebo; Comparison between baseline nail brittleness values and completion values; Test type: Superiority; p = 0.062, t-test, 2 sided — Threshold is p<0.05

5. Secondary Outcome: Number of Days Until the First Nail Chipped
Description: Average number of days post-treatment until the first nail chipped
Time Frame: Baseline to 30 days
Population: - No nail chipping data on 12 participants
Measure: Mean (Standard Deviation); unit: Days
Units Other Than Participants: Hands
Arm/Group | Bimatoprost 0.01% Drops | Placebo
Number analyzed (Participants) | 26 | 26
Number analyzed (Hands) | 26 | 26
Days | 8.38 (9.36) | 6.26 (8.12)

6. Secondary Outcome: Change in Skin Pigmentation on Hands
Description: Photographs taken (knuckle to fingertips over white paper with consistent bulb illumination at the site), with an Apple iPhone 6 (Cupertino, CA, USA) and examined. The investigators reviewed the anonymous photos by number to look for comparative skin pigmentation (increased pigmentation, decreased pigmentation, no change in pigmentation) changes on the hands.
Time Frame: Baseline, 30 days
Population: * Data omitted for 4 subjects with pigmented control and medication hands
  * No data for an additional 4 subjects due to poor photo quality
Measure: Count of Units; unit: Hands
Units Other Than Participants: Hands
Arm/Group | Bimatoprost 0.01% Drops | Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (Hands) | 30 | 30
Hands
  Decreased Pigmentation | 10 | 0
  No Change in Pigmentation | 19 | 30
  Increased Pigmentation | 1 | 0

7. Secondary Outcome: Change in Hirsutism on Hands
Description: Photographs taken (knuckle to fingertips over white paper with consistent bulb illumination at the site), with an Apple iPhone 6 (Cupertino, CA, USA) and examined. The investigators reviewed the anonymous photos by number to look for comparative (increased hair growth, decreased hair growth, no change) hair changes on the hands.
Time Frame: Baseline, 30 days
Population: - No data on 4 participants due to poor photo quality
Measure: Count of Units; unit: Hands
Units Other Than Participants: Hands
Arm/Group | Bimatoprost 0.01% Drops | Placebo
Number analyzed (Participants) | 34 | 34
Number analyzed (Hands) | 34 | 34
Hands
  Decreased Hair Growth | 0 | 0
  No Change in Hair Growth | 34 | 34
  Increased Hair Growth | 0 | 0

ADVERSE EVENTS:
Arm/Group | Bimatoprost 0.01% Drops | Placebo
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 0/38 | 0/38

LIMITATIONS AND CAVEATS:
Nail chipping reduced the N value at the completion of the study. Suggestion is to etch the nail surface to create a mark, then measure from the nail fold to the nail etch at the end of the trial period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes